CLINICAL TRIAL: NCT00162032
Title: A Phase III, Open-Label, Non-Randomized, International, Multicenter Trial to Evaluate the Efficacy and Safety of CARDIOLITE® Myocardial Perfusion Imaging in Pediatric Subjects With Kawasaki Disease
Brief Title: A Study to Evaluate the Use and Safety of CARDIOLITE® in Pediatric Patients With Kawasaki Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARDIOLITE® 301
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children (Ages 4-11) (Other): Children 4-11 years of age, intervention Sestamibi
  Interventions: Drug: Sestamibi
- Adolescents (Ages 12-16) (Other): Adolescents 12-16 years of age, intervention Sestamibi
  Interventions: Drug: Sestamibi

INTERVENTIONS:
Drug: Sestamibi — Sestamibi
  Other Names: Cardiolite

SUMMARY:
Determine the predictive value of CARDIOLITE® rest and stress myocardial perfusion imaging (MPI) to define a pediatric population with Kawasaki Disease (KD) at high and low risk of developing cardiac events.

DETAILED DESCRIPTION:
The purpose of this clinical research study is to determine how well CARDIOLITE® rest and stress myocardial (heart) imaging can define the pediatric Kawasaki disease (KD) population into high and low risk categories of developing cardiac (heart) events (complications) from 1 year through 3 years after image completion. The safety of CARDIOLITE® rest and stress heart imaging will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 4 and 16
* Meet the epidemiological definition of Kawasaki Disease or have a diagnosis of incomplete KD, including evidence of coronary artery disease as determined by their physician.
* Be able to exercise adequately to achieve 85% age predicted maximum heart rate

Exclusion Criteria:

* Terminal illness where expected survival is < 6 months

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 445 (Actual)
Dates: Start 2005-08; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhu, MD,, Study Director — Lantheus Medical Imaging
Locations (49):
- United States (28):
  - Local Institution, Anchorage, Alaska
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Los Angeles, California
  - Local Institution, Orange, California
  - Local Institution, San Diego, California
  - Local Institution, Denver, Colorado
  - Local Institution, Hartford, Connecticut
  - Local Institution, New Haven, Connecticut
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Chicago, Illinois
  - Local Institution, Park Ridge, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Lexington, Kentucky
  - Local Institution, Boston, Massachusetts
  - Local Institution, Las Vegas, Nevada
  - Local Institution, New Hyde Park, New York
  - Local Institution, New York, New York
  - Local Institution, Durham, North Carolina
  - Local Institution, Greenville, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Local Institution, Hershey, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Seattle, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Milwaukee, Wisconsin
- Brazil (5):
  - Local Institution, Belo Horizonte
  - Local Institution, Campinas
  - Local Institution, Curitiba
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (4):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- Local Institution, Quezon City, Philippines
- South Korea (5):
  - Local Institution, Daejeon
  - Local Institution, Pusan
  - Local Insitution, Seoul
  - Local Institution, Suwon
  - Local Institution, Wŏnju
- Taiwan (4):
  - Local Institution, Changhua
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Taipei
- Thailand (2):
  - Local Institution, Bangkok
  - Local Institution, Hat Yai

RESULTS

PARTICIPANT FLOW:
Groups:
- Children (Ages 4-11): Arm A children 4-11 years of age
- Adolescents (Ages 12-16): Arm B children 12-16 years of age
Period: Overall Study
Arm/Group | Children (Ages 4-11) | Adolescents (Ages 12-16)
Started | 329 | 116
Completed | 324 (Completed is all subjects who completed 3 yr FU whether or not they were seen in the previous year.) | 114 (Completed is all subjects who completed 3 yr FU whether or not they were seen in the previous year.)
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 4 | 2
Not completed — Reason not specified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children (Ages 4-11) | Adolescents (Ages 12-16) | Total
Number analyzed (Participants) | 329 | 116 | 445
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 329 | 116 | 445
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (2.16) | 13.6 (1.31) | 9.0 (3.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 40 | 144
  Male | 225 | 76 | 301
Region of Enrollment [Number; unit: participants]
  United States | 64 | 39 | 103
  Philippines | 33 | 8 | 41
  Taiwan | 85 | 27 | 112
  Canada | 18 | 17 | 35
  Brazil | 34 | 5 | 39
  Thailand | 46 | 6 | 52
  Korea, Republic of | 43 | 10 | 53
  Singapore | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Determine the Predictive Value of Cardiolite® Rest and Stress MPI to Define Pediatric Populations With Kawasaki Disease at High and Low Risk of Developing Cardiac Events.
Description: The proportion of all patients who experienced cardiac events among patients with abnormal (SSS >=4, high risk) and normal (SSS <4, low risk) Cardiolite MPI scans during the follow-up period. A log-rank statistic (2-sided, alpha = 0.05) was computed to compare cardiac event-free survival in the high risk and low risk groups. The cardiac event rate is the cumulative event rate based on a Kaplan-Meier estimate conditional on the SPECT MPI score result.
Time Frame: 3 years
Population: Had SPECT Myocardial perfusion imaging tests and experienced a cardiac event
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Children (4 -11 Years) Normal: SSS (summed stress score) <=4, low risk
- Adolescents (12-16 Years) Normal: SSS (summed stress score) <4, low risk
- Children (4-11 Years) Abnormal: SSS (summed stress score)>4, high risk
- Adolescents (12-16 Years) Abnormal: sss (summed stress score >4, high risk
Arm/Group | Children (4 -11 Years) Normal | Adolescents (12-16 Years) Normal | Children (4-11 Years) Abnormal | Adolescents (12-16 Years) Abnormal
Number analyzed (Participants) | 287 | 93 | 26 | 19
proportion of participants | 0.041 [0.015 to 0.066] | 0.033 [0.000 to 0.071] | 0.115 [0.000 to 0.238] | 0.233 [0.000 to 0.493]

2. Secondary Outcome: Estimate the Performance of Cardiolite® Rest and Stress MPI for the Detection of Myocardial Ischemia in Adolescents and Children Versus Coronary Angiography
Description: Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of myocardial perfusion imaging (MPI) for the diagnosis of ischemic heart disease (IHD) relative to coronary angiography. Coronary stenoses of ≥ 50% were classified as disease. SSS > 4 in MPI was classified as positive for IHD.
Time Frame: 6 months
Population: Per-protocol population of pooled adolescents and children who underwent coronary angiography
Measure: Number (95% Confidence Interval); unit: proportion
Groups:
- Angiography Subjects: Subset of pooled adolescent and child subjects who underwent coronary angiography
Arm/Group | Angiography Subjects
Number analyzed (Participants) | 50
proportion
  Sensitivity | 0.35 [0.11 to 0.69]
  Specificity | 0.62 [0.45 to 0.77]
  Positive Predictive Value | 0.21 [0.06 to 0.46]
  Negative Predictive Value | 0.77 [0.59 to 0.90]

3. Secondary Outcome: Incidence of Hard Cardiac Events
Description: Examine the incidence of hard cardiac events (myocardial infarction [MI] or cardiac death) in KD subjects with positive and negative MPI scans.
Time Frame: 3 years
Population: All subjects who had undergone stress cardiac MPI studies
Measure: Number; unit: participants
Arm/Group | Children (4 -11 Years) Normal | Adolescents (12-16 Years) Normal | Children (4-11 Years) Abnormal | Adolescents (12-16 Years) Abnormal
Number analyzed (Participants) | 287 | 93 | 26 | 19
participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Estimate the Performance of Cardiolite® Rest and Stress MPI for the Detection of Myocardial Ischemia in the Left Anterior Descending (LAD) Artery in Adolescents and Children Versus Coronary Angiography
Description: Sensitivity, specificity, PPV, and NPV of SDS for myocardial perfusion corresponding to the left anterior descending (LAD) for the diagnosis of IHD in the distribution of the left anterior descending (LAD) artery relative to coronary angiography based diagnosis were determined. Coronary stenoses of ≥ 50% for arteries associated with LAD territories were classified as LAD disease. SDS LAD > 1 was classified as positive for IHD for the LAD distribution.
Time Frame: 24 hours
Measure: Number (95% Confidence Interval); unit: proportion
Groups:
- Children (Ages 4-11): Arm A children 4-11 years of age who underwent coronary angiography
- Adolescents (Ages 12-16): Arm B adolescents 12-16 years of age who underwent coronary angiography
Arm/Group | Children (Ages 4-11) | Adolescents (Ages 12-16)
Number analyzed (Participants) | 29 | 22
proportion
  Sensitivity | .25 [0.01 to 0.81] | 0.00 [0.00 to 0.71]
  Specificity | 0.76 [0.55 to 0.91] | 0.74 [0.49 to 0.91]
  Positive Predictive Value | 0.14 [0.00 to 0.58] | 0.00 [0.00 to 0.52]
  Negative Predictive Value | 0.86 [0.65 to 0.97] | 0.82 [0.57 to 0.96]

5. Secondary Outcome: Predictive Value of Cardiolite For Cardiac Events
Description: Determine the incidence of cardiac events occurring over a 6 month follow up period in pediatric subjects with normal myocardial perfusion scans.
Time Frame: 6 months
Population: Efficacy Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Children (4 -11 Years) Normal | Adolescents (12-16 Years) Normal | Children (4-11 Years) Abnormal | Adolescents (12-16 Years) Abnormal
Number analyzed (Participants) | 287 | 93 | 26 | 19
Participants | 3 | 1 | 3 | 2

ADVERSE EVENTS:
Time Frame: AEs within 24+- 12 hours. SAEs up to 14 days.
Groups:
- Adolescents (Ages 12-16): Arm B adolescents 12-16 years of age
Arm/Group | Children (Ages 4-11) | Adolescents (Ages 12-16)
Serious Adverse Events (participants affected / at risk) | 1/329 | 0/116
Other Adverse Events (participants affected / at risk) | 8/329 | 5/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children (Ages 4-11) (N=329) | Adolescents (Ages 12-16) (N=116)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Subject 014-006 was a 5-year old white female. The subject received a total dose of Cardiolite on 05 June 2006 of 16.9 mCi. The nuclear medicine technician incorrectly calculated the doses based on a weight of 40 kg rather 40 lbs (18.1 kg).
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children (Ages 4-11) (N=329) | Adolescents (Ages 12-16) (N=116)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
Limited number of subjects receiving coronary angiography limit the clinical implications of this endpoint comparing MPI and coronary angiography in children and adolescents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days